CLINICAL TRIAL: NCT03200574
Title: Behavior of Valve Leaflets and the Incidence of Reduced Mobility Post-surgical Aortic Valve Implant
Brief Title: Behavior of Valve Leaflets Following Aortic Valve Implant
Acronym: BELIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corcym S.r.l (Industry)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR002
Record Dates: First submitted 2017-06-09; First posted 2017-06-27 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Aortic-valve Replacement
Keywords: Perceval

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Aortic Valve (Other): LivaNova bioprosthetic aortic heart valve replacement
  Interventions: Diagnostic Test: 4D Cardiac CT Scan; Device: LivaNova Bioprothetic Aortic Valve Implant

INTERVENTIONS:
Diagnostic Test: 4D Cardiac CT Scan — 4D CT scan obtained at minimum of 1 month after the discontinuation of the anticoagulation or dual antiplatelet therapy
Device: LivaNova Bioprothetic Aortic Valve Implant — Study includes patients that have received the commercially approved LivaNova bioprosthetic aortic heart valve Perceval, as standard of care.

SUMMARY:
This is a prospective, interventional, multi-center trial to report the overall incidence of reduced leaflet motion identified by CT imaging in patients receiving a commercially approved LivaNova bioprosthetic aortic heart valve up to 1 year post implant.

DETAILED DESCRIPTION:
This is a prospective, interventional, multi-center trial to report the overall incidence of reduced leaflet motion identified by CT imaging in patients receiving a commercially approved LivaNova bioprosthetic aortic heart valve up to 1 year post implant, on patients that are off anticoagulation for at least 30 days. A minimum of 75 subjects with evaluable 4D CT scans will be enrolled at approximately 11 investigational sites where the devices are commercially available. For asymptomatic subjects, PIs and subjects will be blinded from the CT imaging results and from the Core Lab findings.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has been successfully implanted with a commercially approved LivaNova bioprosthetic valve according to the instructions for use (IFU)
2. The subject has signed the informed consent.
3. The subject is at least 18 years of age at the time of implant and consent signature
4. The subject will be available for post-operative follow-up through one year

Exclusion Criteria:

1. The subject has a planned concomitant cardiac procedure other than coronary artery bypass graft (CABG) and septal myectomy, including MAZE procedures, atrial fibrillation surgery, and left atrial appendage exclusion or resection, or has a prosthetic heart valve or annuloplasty ring in any position
2. The subject has any medical condition requiring long term (> 6 months) anticoagulation or dual antiplatelet therapy
3. The subject has any clinical condition precluding the use of CT imaging with contrast
4. The subject had a stroke or myocardial infarction (STEMI and NSTEMI) within 30 days of the planned valve implant surgery
5. The subject has active endocarditis, myocarditis, or sepsis
6. The subject is in cardiogenic shock manifested by low cardiac output and needing hemodynamic support
7. The subject is already included in another clinical trial that could confound the results of this clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Washington Adventist Hospital; Federico Asch, MD, Principal Investigator — Medstar Health Research Institute
Locations (11):
- United States (8):
  - St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - Maine Medical Center, Scarborough, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Oakwood Hospital, Dearborn, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Baptist Hospital, St Louis, Missouri
  - Centennial, Nashville, Tennessee
  - Valley Health, Winchester, Virginia
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Universite Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams DH, Popma JJ, Reardon MJ. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 Sep 4;371(10):967-8. doi: 10.1056/NEJMc1408396. No abstract available. PMID 25184874
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Mohr FW, Holzhey D, Mollmann H, Beckmann A, Veit C, Figulla HR, Cremer J, Kuck KH, Lange R, Zahn R, Sack S, Schuler G, Walther T, Beyersdorf F, Bohm M, Heusch G, Funkat AK, Meinertz T, Neumann T, Papoutsis K, Schneider S, Welz A, Hamm CW; GARY Executive Board. The German Aortic Valve Registry: 1-year results from 13,680 patients with aortic valve disease. Eur J Cardiothorac Surg. 2014 Nov;46(5):808-16. doi: 10.1093/ejcts/ezu290. Epub 2014 Jul 30. PMID 25079769
- [Background] Laschinger JC, Wu C, Ibrahim NG, Shuren JE. Reduced Leaflet Motion in Bioprosthetic Aortic Valves--The FDA Perspective. N Engl J Med. 2015 Nov 19;373(21):1996-8. doi: 10.1056/NEJMp1512264. Epub 2015 Oct 5. No abstract available. PMID 26437127
- [Background] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Background] Beholz S, Repossini A, Livi U, Schepens M, El Gabry M, Matschke K, Trivedi U, Eckel L, Dapunt O, Zamorano JL. The Freedom SOLO valve for aortic valve replacement: clinical and hemodynamic results from a prospective multicenter trial. J Heart Valve Dis. 2010 Jan;19(1):115-23. PMID 20329497
- [Background] Thalmann M, Grubitzsch H, Matschke K, Glauber M, Tan E, Francois K, Amorim MJ, Hensens AG, Cesari F, Feyrer R, Diegeler A, Veit F, Repossini A; Freedom Solo Investigators. A European Multicenter Study of 616 Patients Receiving the Freedom Solo Stentless Bioprosthesis. Ann Thorac Surg. 2016 Jan;101(1):100-8. doi: 10.1016/j.athoracsur.2015.06.096. Epub 2015 Oct 9. PMID 26443880
- [Background] Grubitzsch H, Wang S, Matschke K, Glauber M, Heimansohn D, Tan E, Francois K, Thalmann M. Clinical and haemodynamic outcomes in 804 patients receiving the Freedom SOLO stentless aortic valve: results from an international prospective multicentre study. Eur J Cardiothorac Surg. 2015 Mar;47(3):e97-104. doi: 10.1093/ejcts/ezu471. Epub 2014 Dec 13. PMID 25501554
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):e57-185. doi: 10.1016/j.jacc.2014.02.536. Epub 2014 Mar 3. No abstract available. PMID 24603191
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 88 subjects undergoing AVR with the commercially available Perceval S Valve (Manufacturer Livanova, now transitioned to Corcym), having signed informed consent and willing and able to undergo 4D CT assessments with contrast (or alternatively TEE) were enrolled in the study. The study was forseeing 24 month of enrollment and 1 Year follow-up. The first enrolment occured on on August 12, 2017, and the last enrollment on May 22, 2019 in a total of 10 clinical study sites.
Period: Overall Study
Arm/Group | Aortic Valve
Started | 88 (96 patients were consented, 8 not eligible and 88 enrolled)
Completed | 71
Not Completed | 17
Not completed — Death | 4
Not completed — Withdrawal by Subject | 8
Not completed — Long-Term need for anticoagulation | 1
Not completed — Relocation | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 78
  More than one race | 3
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Leaflet Motion
Description: Report the overall incidence of reduced leaflet motion identified by CT imaging in commercially approved LivaNova bioprosthetic aortic heart valves up to 1 year post implant on patients that are off anticoagulation for at least 30 days.
  The valve leaflets will be assessed using 4D-VR (volume-rendered) CT imaging. Leaflet motion in all leaflets will be defined as normal, mildly reduced (<50% reduction in leaflet opening), moderately reduced (50-70% reduction in leaflet motion), severely reduced (>70% reduction in leaflet motion) and immobile (no or negligible leaflet motion).
Time Frame: 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 12

2. Secondary Outcome: Leaflet Motion in Symptomatic and Asymptomatic Subjects Outcomes
Description: Incidence of reduced leaflet motion in symptomatic and asymptomatic subjects based on CT outcomes and anticoagulation and dual antiplatelet treatment modalities up to 1 year post-implant.
  The valve leaflets will be assessed using 4D-VR (volume-rendered) CT imaging. Leaflet motion in all leaflets will be defined as normal, mildly reduced (<50% reduction in leaflet opening), moderately reduced (50-70% reduction in leaflet motion), severely reduced (>70% reduction in leaflet motion) and immobile (no or negligible leaflet motion).
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Groups:
- Asymptomatic Patients; Symtomatic Patients: LivaNova bioprosthetic aortic heart valve replacement
  4D Cardiac CT Scan: 4D CT scan obtained at minimum of 1 month after the discontinuation of the anticoagulation or dual antiplatelet therapy
  LivaNova Bioprothetic Aortic Valve Implant: Study includes patients that have received the commercially approved LivaNova bioprosthetic aortic heart valve Perceval, as standard of care.
Arm/Group | Asymptomatic Patients | Symtomatic Patients
Number analyzed (Participants) | 87 | 1
Participants | 11 | 1

3. Secondary Outcome: Reduced Leaflet Motion Through 4D Volume-rendered CT Scan
Description: Incidence of reduced leaflet motion through 4D volume-rendered CT scan with contrast up to 1 year post-implant, in subjects in which reduced leaflet motion was previously detected.
  The valve leaflets will be assessed using 4D-VR (volume-rendered) CT imaging. Leaflet motion in all leaflets will be defined as normal, mildly reduced (<50% reduction in leaflet opening), moderately reduced (50-70% reduction in leaflet motion), severely reduced (>70% reduction in leaflet motion) and immobile (no or negligible leaflet motion).
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Reduction in Leaflet Motion by Relationship to Devices or Procedure
Description: Incidence of reduced leaflet motion considering relationship to the devices, procedure, or other causes up to 1 year post-implant The valve leaflets will be assessed using 4D-VR (volume-rendered) CT imaging. Leaflet motion in all leaflets will be defined as normal, mildly reduced (<50% reduction in leaflet opening), moderately reduced (50-70% reduction in leaflet motion), severely reduced (>70% reduction in leaflet motion) and immobile (no or negligible leaflet motion).
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Reduced Leaflet Motion (RLM) Overall: LivaNova bioprosthetic aortic heart valve replacement
  4D Cardiac CT Scan: 4D CT scan obtained at minimum of 1 month after the discontinuation of the anticoagulation or dual antiplatelet therapy
  LivaNova Bioprothetic Aortic Valve Implant: Study includes patients that have received the commercially approved LivaNova bioprosthetic aortic heart valve Perceval, as standard of care.
- Subjects Implanted With Perceval Size S: Subjects with RLM implanted with Perceval size S
- Subjects Implanted With Perceval S Size M: Subjects with RLM implanted with Perceval size M
- Subjects Implanted With Perceval S Size L: Subjects with RLM implanted with Perceval size L
- Subjects Implanted With Perceval Size XL: Subjects with RLM implanted with Perceval size XL
- Subjects Implanted With Perceval Via Minimally Invasive Surgical Approach: Subjects with RML implanted with Perceval via minimally invasive surgical approach
- Subjects Implanted With Perceval Via Full Sternotomy Surgical Approach: Subjects with RLM implanted with Perceval via full sternotomy surgical approach
Arm/Group | Subjects With Reduced Leaflet Motion (RLM) Overall | Subjects Implanted With Perceval Size S | Subjects Implanted With Perceval S Size M | Subjects Implanted With Perceval S Size L | Subjects Implanted With Perceval Size XL | Subjects Implanted With Perceval Via Minimally Invasive Surgical Approach | Subjects Implanted With Perceval Via Full Sternotomy Surgical Approach
Number analyzed (Participants) | 88 | 15 | 19 | 26 | 28 | 41 | 47
Participants | 12 | 1 | 3 | 4 | 4 | 5 | 7

5. Secondary Outcome: Freedom From All-cause Mortality
Description: Number and incidence of subjects free from all-cause mortality
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 84

6. Secondary Outcome: Freedom From Valve Re-intervention
Description: Number and incidence of subjects free from valve reintervention
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 88

7. Secondary Outcome: Freedom From Myocardial Infarction
Description: Number and incidence of subjects free from myocardial infarction
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 88

8. Secondary Outcome: Freedom From Structural Valve Deterioration
Description: Number and incidence of subjects free from structural valve deterioration
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 88

9. Secondary Outcome: Freedom From Moderate or Severe Valve Regurgitation
Description: Number and incidence of subjects free from moderate or severe valve regurgitation
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 88

10. Secondary Outcome: Freedom From Valve Endocarditis
Description: Number and incidence of subjects free from valve endocarditis
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 88

11. Secondary Outcome: Freedom From Valve Thrombosis
Description: Number and incidence of subjects free from valve thrombosis
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 87

12. Secondary Outcome: Freedom From Thromboembolic Events
Description: Number and incidence of subjects free from thromboembolic events
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 82

13. Secondary Outcome: Freedom From Hemolysis
Description: Number and incidence of subjects free from hemolysis
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 88

14. Secondary Outcome: Freedom From Major Bleeding
Description: Number and incidence of subjects free from major bleeding
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 88
Participants | 85

15. Secondary Outcome: New York Heart Association (NYHA) Assessment
Description: Number and incidence of subjects in the different NYHA class at 1 year post-implant.
  NYHA I = Subjects with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or angina.
  NYHA II = Subjects with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or angina.
  NYHA III = Subjects with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or angina.
  NYHA IV = Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or angina may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 69
Participants
  NYHA class I | 52
  NYHA class II | 17
  NYHA Class III | 0
  NYHA class IV | 0

16. Secondary Outcome: Aortic Peak Gradient Through Transthoracic Echocardiogram (TTE)
Description: Summary statistics (means, Standard Deviation, median, quartiles and range values for continuous variables; count and frequency distributions for categorical variables) of Hemodynamic assessment up to 1 year post-implant through Echocardiographic Core Lab transthoracic echocardiogram (TTE)
Time Frame: up to 1 year post-implant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Valve
Number analyzed (Participants) | 68
mmHg | 22.6 (9.6)

17. Secondary Outcome: Aortic Mean Gradient Through Transthoracic Echocardiogram (TTE)
Description: as for outcome 16
Time Frame: up to 1 year post-implant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Valve
Number analyzed (Participants) | 68
mmHg | 12.5 (5.9)

18. Secondary Outcome: Effective Orifice Area Through Transthoracic Echocardiogram (TTE)
Description: as for outcome 16
Time Frame: up to 1 year post-implant
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Aortic Valve
Number analyzed (Participants) | 68
cm2 | 1.7 (0.5)

19. Secondary Outcome: Global Aortic Regurgitation Through Transthoracic Echocardiogram (TTE)
Description: as for outcome 16
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 68
Participants
  No regurgitation | 51
  Trace | 4
  Mild | 9
  Moderate | 1
  Not evaluable | 3

20. Secondary Outcome: Central Aortic Regurgitation Through Transthoracic Echocardiogram (TTE)
Description: as for outcome 16
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 68
Participants
  None | 60
  Trace | 2
  Mild | 5
  Not evaluable | 1

21. Secondary Outcome: Paravalvular Aortic Regurgitation Through Transthoracic Echocardiogram (TTE)
Description: as for outcome 16
Time Frame: up to 1 year post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve
Number analyzed (Participants) | 68
Participants
  None | 60
  Trace | 1
  Mild | 6
  Not evaluable | 1

ADVERSE EVENTS:
Time Frame: Overall incidences of Serious Adverse Events reported between implant (day 0) and 1 year follow up
Description: The investigators were required to report only SAEs to the Sponsor defined as Adverse event that led to any of the following
  1. death,
  2. serious deterioration in the health of the subject, users, or other persons
  3. foetal distress, foetal death, a congenital abnormality, or birth defect including physical or mental impairment.
  Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Aortic Valve
All-Cause Mortality (participants affected / at risk) | 4/88
Serious Adverse Events (participants affected / at risk) | 38/88
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Valve (N=88)
Access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Bleeding disorders (Blood and lymphatic system disorders) | 3 (3)
Blood disorders (Blood and lymphatic system disorders) | 2 (2)
Arrhythmias and conduction disorders (Cardiac disorders) | 12 (12)
Cardiac arrest/cardiorespiratory arrest (Cardiac disorders) | 1 (1) — leading to death
Cardiac decompensation (Cardiac disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Thrombosis, Valve (Cardiac disorders) | 1 (1)
Gastrointestinal and hepatobiliary disorders (Gastrointestinal disorders) | 2 (2)
Chest pain, noncardiac (General disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Lab Test abnormality (Investigations) | 1 (1)
Injuries, Trauma, Social circumstances (Social circumstances) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Confusion, Delirium (Nervous system disorders) | 2 (2)
Dizziness / Vertigo (Nervous system disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Other Neurologic Disorder (Nervous system disorders) | 1 (1)
Stroke (CVA) (Nervous system disorders) | 5 (5) — 1 case of Stroke led to death
Syncope / loss of consciousness (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Other renal and genitourinary disorders (Renal and urinary disorders) | 2 (2)
Dyspnoea/Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — leading to death
Arterial stenosis (Vascular disorders) | 1 (1)
Embolization (air, tissue, septic, device) (Vascular disorders) | 2 (2)
Peripheral artery stenosis/peripheral vaso-occlusive disease/peripheral vascular disease (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 4 (4)
Thrombosis, deep vein (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Access site infection (Injury, poisoning and procedural complications) | 1 (1)
Other access site complications (Injury, poisoning and procedural complications) | 1 (1)
Other cardiac disorder (Cardiac disorders) | 1 (1)
Death unknown cause (General disorders) | 1 (1)
Other general system disorders (General disorders) | 1 (1)
Genitourinary infections (Infections and infestations) | 2 (2)
Respiratory system infections (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Skin and subcutaneous infections (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03200574/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT03200574/SAP_001.pdf